CLINICAL TRIAL: NCT00815984
Title: FeNO Result Prediction Factors in Children With Allergic Diseases
Brief Title: Fractional Exhaled Nitric Oxide (FeNO) Result Prediction Factors in Children With Allergic Diseases
Status: Completed | Type: Observational
Sponsor: Medical University of Lodz (Other)
Responsible Party: Iwona Stelmach MD, PhD, Prof, Department of Pediatrics and Allergy, N. Copernicus Hospital, Lodz, Poland
Other Study IDs: RNN/135/08/KE
Record Dates: First submitted 2008-12-30; First posted 2008-12-31 (Estimated); Last update posted 2010-02-10 (Estimated); Status verified 2010-02

CONDITIONS: Asthma; Allergic Rhinitis; Atopic Dermatitis
Keywords: Asthma; Allergic Rhinitis; Atopic Dermatitis; Children; lung function; skin prick tests; FeNO
MeSH Terms: conditions — Asthma; Rhinitis, Allergic; Dermatitis, Atopic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Schoolchildren with asthma.: Schoolchildren with asthma.
  Interventions: Procedure: measurements of lung function tests

INTERVENTIONS:
Procedure: measurements of lung function tests — Measurement of the concentration of FeNO , measurement of spirometry, plethysmography, exercise challenge test (ECT -spirometric), bronchial obstruction reversibility pharmacological test
  Other Names: NO analyzer- Sievers 280i analyzer; Spirometry and Plethysmography - Jaeger; Exercise provocation test treadmill- Kettler

SUMMARY:
In about 800 children with allergic diseases (asthma, allergic rhinitis, atopic dermatitis) the investigators will retrospectively and cross-sectionally analyze the influence/correlation of diagnosis, treatment methods, allergy status (skin prick test results), lung function tests results on/with the concentration of nitric oxide in exhaled breath.

DETAILED DESCRIPTION:
In about 800 children with allergic diseases from our Outpatient Clinic (asthma, allergic rhinitis, atopic dermatitis) we will retrospectively and cross-sectionally analyse the influence/correlation of diagnosis, treatment methods, allergy status (skin prick test results), lung function tests results on/with the concentration of nitric oxide in exhaled breath.

ELIGIBILITY:
Inclusion Criteria:

* Children with asthma (allergic), and/or allergic rhinitis and/or atopic dermatitis

Exclusion Criteria:

* Other chronic diseases
* Asthma exacerbation
* Pregnancy

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children with asthma (allergic), and/or allergic rhinitis and/or atopic dermatitis
Sampling Method: Probability Sample
Enrollment: 800 (Actual)
Dates: Start 2009-01; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Concentration of nitric oxide in exhaled breath. | 1-4 months

CONTACTS AND LOCATIONS:
Overall Officials: Iwona Stelmach, MD PhD Prof, Study Chair — Department of Pediatrics and Allergy, N. Copernicus Hospital, Lodz, Poland; Tomasz Grzelewski, MD, PhD, Principal Investigator — Department of Pediatrics and Allergy, N. Copernicus Hospital, Lodz, Poland
Locations (1):
- Department of Pediatrics and Allergy, N. Copernicus Hospital, Lodz, Poland

REFERENCES:
- [Derived] Grzelewski T, Majak P, Jerzynska J, Stelmach W, Stelmach R, Janas A, Grzelewska A, Witkowski K, Makandjou-Ola E, Stelmach I. The interpretation of exhaled nitric oxide values in children with asthma depends on the degree of bronchoconstriction and the levels of asthma severity. Respir Care. 2014 Sep;59(9):1404-11. doi: 10.4187/respcare.02889. Epub 2013 Dec 31. PMID 24381190